CLINICAL TRIAL: NCT01300338
Title: Does Home Telemonitoring Increase the Number of Diabetic Patients at Goal Blood Pressure in a Primary Care Practice?
Brief Title: Blood Pressure Telemonitoring and Goal Blood Pressure in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Frederick North, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-003562
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Blood Pressure Monitors; Telemetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood pressure with telemetry (Experimental): Home blood pressure monitor with telemetry
  Interventions: Device: Blood pressure monitor with telemetry
- Blood pressure without telemetry (Active Comparator): Home blood pressure self monitor without telemetry.
  Interventions: Device: Home blood pressure monitor without telemetry

INTERVENTIONS:
Device: Blood pressure monitor with telemetry — Blood pressure monitor for home use with readings uploaded to a web server viewable by the diabetes care manager
  Other Names: Ideal Life Blood Pressure Monitor
  Arms: Blood pressure with telemetry
Device: Home blood pressure monitor without telemetry — Self monitor of blood pressure without telemetry
  Other Names: Omron blood pressure monitor
  Arms: Blood pressure without telemetry

SUMMARY:
Does home telemonitoring increase the number of diabetes patients at goal blood pressure in a primary care practice?

DETAILED DESCRIPTION:
This is a randomized control trial, two arms with block randomization. Primary care patients with diabetes and elevated blood pressure randomized to intervention or control. Intervention arm: home telemonitoring using the Ideal Life blood pressure cuff and telephone or internet transmission device to transmit blood pressure information to the Primary care manager team with otherwise normal care manager care. Control arm: Omron (off the shelf) home blood pressure monitor (no transmission of data) and usual care. We will be comparing blood pressure control between groups and provider contacts.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75 (inclusive
* Blood pressure in hypertensive range (systolic >= 140 or diastolic >=90
* Diabetes

Exclusion criteria:

* Pregnancy
* Lack of computer with internet access or phone line
* Lack of English language literacy
* Arm size to large or small for cuff

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick North, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled at the Mayo Clinic in Rochester, Minnesota from March 2011 to October 2012.
Groups:
- Blood Pressure With Telemetry: Blood pressure monitor with telemetry
  blood pressure with telemetry: Blood pressure monitor for home use with readings uploaded to a web server viewable by the diabetes care manager
- Blood Pressure Without Telemetry: Blood pressure self monitor without telemetry
  Home blood pressure monitor without telemetry: Self monitor of blood pressure without telemetry.
Period: Overall Study
Arm/Group | Blood Pressure With Telemetry | Blood Pressure Without Telemetry
Started | 25 | 25
Completed | 20 | 25
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Pressure With Telemetry | Blood Pressure Without Telemetry | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is indicated in years
  years | 63.24 (7.93) | 62.36 (8.55) | 62.8 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Systolic Blood Pressure
Description: Average change in systolic blood pressure (top number of blood pressure reading) from baseline to 6 months.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: Millimeters of Mercury
Arm/Group | Blood Pressure With Telemetry | Blood Pressure Without Telemetry
Number analyzed (Participants) | 20 | 25
Millimeters of Mercury | -3.08 [-8.6 to 2.4] | 2.72 [-5.6 to 11.0]

2. Primary Outcome: Mean Change in Diastolic Blood Pressure
Description: Average change in diastolic blood pressure (bottom number of blood pressure reading) from baseline to 6 months.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: Millimeters of Mercury
Arm/Group | Blood Pressure With Telemetry | Blood Pressure Without Telemetry
Number analyzed (Participants) | 20 | 25
Millimeters of Mercury | -1.92 [-5.2 to 1.4] | 1.72 [-2.3 to 5.7]

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | Blood Pressure With Telemetry | Blood Pressure Without Telemetry
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No